CLINICAL TRIAL: NCT01597570
Title: Clinical Evaluation of Effectiveness and Safety Confirmation Between FASTSEAL® Bioabsorbable Vascular Access Closure System and Perclose® ProGlide Suture-Mediated Closure System; Randomized, Comparative Study
Brief Title: Effectiveness and Safety Confirmation Between FASTSEAL® Bioabsorbable VCD and Perclose® ProGlide SMC System
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Taewoong Medical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FASTSEAL® VCD
Record Dates: First submitted 2012-05-10; First posted 2012-05-14 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: The Patients Who Needed Hemostasis at the Puncture Site of Common Femoral Artety(CFA) Caused by Femoral Angiogram or Intervention After the Catheter Removal
MeSH Terms: interventions — Vascular Closure Devices

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- FASTSEAL® Bioabsorbable VCD (Experimental): Fastseal® Bioabsorbable Vascular Access Closure System
  Interventions: Device: Vascular Closure Device
- Perclose® ProGlide SMC System (Active Comparator): Perclose® ProGlide Suture-Mediated Closure System
  Interventions: Device: Vascular Closure Device

INTERVENTIONS:
Device: Vascular Closure Device — To reduce the TTH(Time to hemostasis) and TTA(Time to ambulation)of common femoral artery(CFA) puncture site
  Other Names: FASTSEAL® Bioabsorbable Vascular Access Closure System /; Perclose® ProGlide Suture-Mediated Closure System

SUMMARY:
It is purposed to verify a superiority of the Fastseal® Bioabsorbable Vascular Access Closure System through effectiveness and safety confirmation of hemostasis (TTH; Time to hemstasis) and ambulation (TTA; Time to ambulation) at the puncture site of common femoral artery (CFA) after the procedures of Fastseal® Biosorbable Vascular Access Closure System or Perclose® ProGlide Suture-Mediated Closure System during 1 month observation.

DETAILED DESCRIPTION:
Prospective, Single blind, randomized

Comparative study using the Fastseal® Bioabsorbable Vascular Access Closure System as an investigational device and the Perclose® ProGlide Suture-Mediated Closure System as a comparator.

After going through the confirmation of inclusion/exclusion criteria with signed subjects, they will have a procedure either of the two devices. The subjects should follow designated physician's instructions accurately during the clinical trial period.There are about 6 times evaluations Including screening.

ELIGIBILITY:
Inclusion Criteria:

* Between 20 years old and 85 years old, randomized
* Patient who submitted a written informed consent for the this trial
* The subjects should be scheduled to have an angiography or intervention through the common femoral artery (CFA).
* The subjects must be used a 6Fr sheath of the Terumo's RadiFocus Introducer II.

Exclusion Criteria:

* In case of the subject has a functure site in both legs.
* The patient who had the closing device insertion or manual compression at the targeted femoral artery within 30 days
* Patients with severe bleeding disorders (Severe bleeding history, blood coagulation disorder, thrombocytopenia (under 100,000 of platelet count), hemophilia, anemia (Hgb<10g/dL, Hct<30%), Thrombasthenia, any related bleeding disorder
* Hypertension patient BP ≥180/110mmHg
* In case of thrombolysis(ex: streptokinase, urokinase, t-PA) within 24hr
* If there is any hematoma, arteriovenous fistula(AVF), false aneurysm existed at the access site of femoral artery
* Severe obesity BMI > 40kg/m2
* In case of prior stent placement or artificial vessel insertion in the common femoral artery(CFA)
* Under 5mm of Common femoral artery (CFA) diameter

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-05; Primary Completion 2012-12-10 (Actual); Study Completion 2012-12-10 (Actual)

PRIMARY OUTCOMES:
TTH; Time to hemostasis | From the procedure start - 1m 30s, 2m 30s, 3m 30s, 4m 30s, 6m 30s, 8m 30s, 10m 30s
  Time interval between procedure and hemostasis

SECONDARY OUTCOMES:
TTA(Time to ambulation) & Failure rate of hemostasis | From the procedure start - 2hr, 4hr, 6hr, 8hr, 12hr
  Time interval between procedure and ambulation

CONTACTS AND LOCATIONS:
Overall Officials: Dongik Kim, Professor Dr., Principal Investigator — Severance Hospital / Radiology
Locations (2):
- South Korea (2):
  - Samsung Medical Center, Seoul, Irwon-Dong, Gangnam-Gu
  - Severance Hospital, Seoul, Seodaemun Gu